CLINICAL TRIAL: NCT00603304
Title: Complementary and Alternative Medicine for Urological Symptoms (CAMUS)
Brief Title: Complementary and Alternative Medicine for Urological Symptoms(CAMUS)
Acronym: CAMUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Office of Dietary Supplements (ODS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Cornell University (Other); New York University (Other); Kaiser Permanente (Other); Northwestern University (Other); Queen's University (Other); University of Colorado, Denver (Other); University of Iowa (Other); University of Maryland (Other); University of Texas (Other); Washington University School of Medicine (Other); Yale University (Other)
Responsible Party: Principal Investigator, Alan Cantor, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X021004002; U01DK063788 (NIH); Tracking # (UAB) 000175609 (Other: Institutional Tracking number for OGCA); NCT00097136 (obsolete NCT alias)
Record Dates: First submitted 2007-12-20; First posted 2008-01-29 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Urological
Keywords: Serenoa repens; Urological symptoms; hyperplasia; BPH
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will take one 320 mg placebo gelcap daily for 24 weeks one gelcap); followed by 640 mg daily for 24 weeks (two gelcaps) followed by 960 mg daily for 24 weeks (three gelcaps).
  Interventions: Drug: Placebo - first 24 weeks; Drug: Placebo - weeks 24 - 48; Drug: Placebo - weeks 48 - 72
- Saw Palmetto (Active Comparator): Extract of Serenoa Repens 320 mg once daily for 24 weeks (one gelcap); followed by 640 mg daily for 24 weeks (two gelcaps) followed by 960 mg daily for 24 weeks (three gelcaps).
  Interventions: Drug: Saw Palmetto - first 24 weeks; Drug: Saw Palmetto - weeks 24 - 48; Drug: Saw Palmetto - weeks 48 - 72

INTERVENTIONS:
Drug: Saw Palmetto - first 24 weeks — Participants will take one 320 mg chocolate-colored soft gelcaps containing a standardized saw palmetto fruit extract for 24 weeks.
  Arms: Saw Palmetto
Drug: Placebo - first 24 weeks — Participants will take one 320 mg chocolate-colored soft gelcaps containing a placebo for 24 weeks.
  Arms: Placebo
Drug: Saw Palmetto - weeks 24 - 48 — Participants will take 640 mg (2) chocolate-colored soft gelcaps containing a standardized saw palmetto fruit extract for 24 weeks.
  Arms: Saw Palmetto
Drug: Placebo - weeks 24 - 48 — Participants will take 640 mg (2) chocolate-colored soft gelcaps containing a placebo for 24 weeks.
  Arms: Placebo
Drug: Saw Palmetto - weeks 48 - 72 — Participants will take 960 (3) mg chocolate-colored soft gelcaps containing a standardized saw palmetto fruit extract for 24 weeks.
  Arms: Saw Palmetto
Drug: Placebo - weeks 48 - 72 — Participants will take 960 (3) mg chocolate-colored soft gelcaps containing a placebo for 24 weeks.
  Arms: Placebo

SUMMARY:
The CAMUS trial will test Saw palmetto in about 369 men. Men who decide to be part of the CAMUS trial will be given one out of two possible treatments at random. One out of every two men would get an inactive placebo treatment. One out of every two men would get Saw palmetto pills.

This kind of scientific study is the best way to find out if the plant extracts really work to prevent men with benign prostatic hyperplasia (BPH) from getting worse. During the study, men will not know which of the two treatments they are assigned to. They will be followed very closely by a study team every 12 weeks to see how they are doing. Men in the CAMUS trial will be studied over 72 weeks. Tests and all medications needed as part of the study will be provided at no charge to the participant. Participants will be responsible for all other costs not associated with the study tests and medications. All information on study participants will be held in the strictest confidence and no one would have access to patient information other than the required authorized health care and research personnel.

DETAILED DESCRIPTION:
The CAMUS trial is studying the outcomes using herbal therapy for benign prostatic hyperplasia (BPH).

BPH is a common problem for older men. With BPH, the prostate grows larger. Over time, this growth can cause bothersome urinary symptoms. These symptoms can include frequent and/or urgent urination during the day or at night. Men with BPH can also have a weak urine stream, a stream that stops and starts, a feeling of not emptying the bladder all the way, and/or a need to strain to get urination started. BPH is NOT the same as prostate cancer.

A number of natural products (extracts of different plants) seem to be able to reduce the bothersome symptoms of BPH with very few side effects over a few months. One of the plant extracts comes from the dwarf palm tree (Saw palmetto). The investigators do not know whether these plant extracts will reduce the symptoms of BPH over a longer period of treatment.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, potential participants must meet all of the following eligibility criteria:

1. Male at least 45 years of age.
2. Peak urinary flow rate at least 4 ml/sec with a voided volume of at least 125 ml.
3. AUA symptom score ≥ 8 and ≤ 24 at both screening visits.
4. Voluntarily signed informed consent agreement prior to the performance of any study procedures.

Exclusion Criteria:

Potential participants that meet any of the following exclusion criteria will be excluded from the full-scale trial:

1. Any prior invasive intervention for BPH.
2. Phytotherapy for BPH or a 5-alpha reductase inhibitor within 3 months.
3. Alpha blocker within one month.
4. Reported allergic reaction to Serenoa repens.
5. Taken phenylephrine, pseudoephedrine, tricyclic antidepressants, and anticholinergic or cholinergic medication within 4 weeks of the first screening visit, with the following exception: topical anticholinergic eye drops used for glaucoma.
6. Taken an estrogen, androgen, or any drug producing androgen suppression, or anabolic steroids within 6 months.
7. Known clinically significant renal impairment (i.e., creatinine greater than 2.0 mg/dl).
8. Alanine aminotransferase(ALT)serum glutamic pyruvic transaminase(SGPT), aspartate aminotransferase(AST)serum glutamic oxaloacetic transaminase (SGOT) or gamma-glutamyltranspeptidase (GGT) value greater than 3 times the upper limit of normal in the clinical center lab at SV1.0; confirmed on a second measurement.
9. Prothrombin time greater than 3 seconds above the upper limit of normal, or more than 3 seconds above the control value in the clinical center at SV1.0; confirmed on a second measurement.
10. Electrocardiogram (ECG) reading at the clinical center at SV1.0 suggesting active ischemia or recent myocardial infarction until appropriate consultation confirms the absence of an acute coronary syndrome.
11. Prostate-specific antigen (PSA) level greater than 10 ng/ml at the first screening visit.
12. Requires the daily use of a pad or device for incontinence, or International Continence Society male incontinence symptom (ICSmaleIS) score >14 at screening.
13. Unstable medical condition within the past 3 months.
14. History or current evidence of carcinoma of the prostate or bladder, pelvic radiation or surgery, urethral stricture, or prior surgery for bladder neck obstruction.
15. Active urinary tract disease or has undergone cystoscopy or biopsy of the prostate within one month prior to the first screening visit or has an imminent need for urologic surgery.
16. Known primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function.
17. Documented bacterial prostatitis within the past year.
18. Two documented independent urinary tract infections of any type in the past year.
19. Known severe bleeding disorder or need for ongoing therapeutic anticoagulation with coumadin or heparin.
20. Cancer, which is not considered cured (except basal cell or squamous cell carcinoma of the skin). A potential participant is considered cured if there has been no evidence of cancer within five years of randomization. A history of bladder cancer or prostate cancer is exclusionary whether the participant is considered cured or not.
21. Unable to follow protocol directions due to organic brain or psychiatric disease.
22. History of alcoholism or any other substance abuse, which, in the opinion of the investigator, would affect compliance with the protocol.
23. Any serious medical condition likely to impede successful completion of the study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Barry, MD, Study Chair — Massachusetts General Hospital; Alan Cantor, PhD, Principal Investigator — The University of Alabama at Birmingham
Locations (11):
- United States (10):
  - Kaiser Permanente Division of Research, Oakland, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - New York University, New York, New York
  - Cornell University, New York, New York
  - University of Texas - Southwestern Medical Center, Dallas, Texas
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Background] Lee J, Andriole G, Avins A, Crawford ED, Foster H, Kaplan S, Kreder K, Kusek J, McCullough A, McVary K, Meleth S, Naslund M, Nickel JC, Nyberg L, Roehrborn C, Dale Williams O, Barry M. Redesigning a large-scale clinical trial in response to negative external trial results: the CAMUS study of phytotherapy for benign prostatic hyperplasia. Clin Trials. 2009 Dec;6(6):628-36. doi: 10.1177/1740774509352199. Epub 2009 Dec 9. PMID 20007408
- [Background] Lee JY, Foster HE Jr, McVary KT, Meleth S, Stavris K, Downey J, Kusek JW. Recruitment of participants to a clinical trial of botanical therapy for benign prostatic hyperplasia. J Altern Complement Med. 2011 May;17(5):469-72. doi: 10.1089/acm.2010.0300. Epub 2011 May 9. PMID 21554128
- [Result] Barry MJ, Avins AL, Meleth S; Complementary and Alternative Medicine for Urological Symptoms Study Group. Performance of the American Urological Association Symptom Index with and without an additional urge incontinence item. Urology. 2011 Sep;78(3):550-4. doi: 10.1016/j.urology.2011.04.017. Epub 2011 Jul 8. PMID 21741692
- [Result] Helfand BT, McVary KT, Meleth S, Sharp V, Foster H, Naslund M, Williams OD; CAMUS Study Group. The relationship between lower urinary tract symptom severity and sleep disturbance in the CAMUS trial. J Urol. 2011 Jun;185(6):2223-8. doi: 10.1016/j.juro.2011.02.012. Epub 2011 Apr 17. PMID 21497839
- [Result] Barry MJ, Meleth S, Lee JY, Kreder KJ, Avins AL, Nickel JC, Roehrborn CG, Crawford ED, Foster HE Jr, Kaplan SA, McCullough A, Andriole GL, Naslund MJ, Williams OD, Kusek JW, Meyers CM, Betz JM, Cantor A, McVary KT; Complementary and Alternative Medicine for Urological Symptoms (CAMUS) Study Group. Effect of increasing doses of saw palmetto extract on lower urinary tract symptoms: a randomized trial. JAMA. 2011 Sep 28;306(12):1344-51. doi: 10.1001/jama.2011.1364. PMID 21954478
- [Derived] Helfand BT, Lee JY, Sharp V, Foster H, Naslund M, Williams OD, McVary KT; CAMUS Study Group. Associations between improvements in lower urinary tract symptoms and sleep disturbance over time in the CAMUS trial. J Urol. 2012 Dec;188(6):2288-93. doi: 10.1016/j.juro.2012.07.104. Epub 2012 Oct 22. PMID 23083656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1032 men were prescreened for Complementary and Alternative Medicine for Urological Symptoms (CAMUS), usually by telephone; interested and preliminary eligible men were scheduled for a first screening visit.
Groups:
- Saw Palmetto: Participants received one, two, and then three 320 mg chocolate-colored soft gelcaps containing a standardized saw palmetto fruit extract with dose escalations at 24 and 48 weeks.
- Placebo: Participants received either one, two, and then three 320 mg chocolate-colored placebo gelcaps with dose escalations at 24 and 48 weeks.
Period: Overall Study
Arm/Group | Saw Palmetto | Placebo
Started | 183 | 186
Completed | 151 | 155
Not Completed | 32 | 31
Not completed — Lost to Follow-up | 5 | 7
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 4 | 2
Not completed — Unacceptable Treatment Toxicity | 5 | 8
Not completed — Crossed Over to Open Label Therapy | 3 | 3
Not completed — Exclusionary Medication | 2 | 3
Not completed — Non-Compliant | 0 | 1
Not completed — Moved Away | 0 | 2
Not completed — Other | 2 | 0
Not completed — Patient Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saw Palmetto | Placebo | Total
Number analyzed (Participants) | 183 | 186 | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 123 | 125 | 248
  >=65 years | 60 | 61 | 121
Age Continuous [Mean (Standard Deviation); unit: years] | 61.25 (8.72) | 60.70 (8.08) | 60.86 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 183 | 186 | 369
Region of Enrollment [Number; unit: participants]
  United States | 167 | 169 | 336
  Canada | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mean and Standard Deviation of the Participant American Urological Association (AUA)Symptom Score Between Baseline and Week 72 for CAMUS Participants.
Description: The primary outcome was the mean difference in the AUA Symptom Score between baseline and 72 weeks between the saw palmetto and placebo groups. The AUA Symptom Score index is a seven item questionnaire assessing the frequency of lower urinary tract symptoms (LUTS). The questions are scored on a scale of zero to five, with zero being never, one to four being one to four accordingly, and five equaling five or more times. A Symptom Index is determined by adding the scores. The lowest possible score is 0 and the highest possible score is 35, which would represent the highest level of pain and discomfort.
Time Frame: Baseline to 72 weeks
Population: The primary analysis was a modified intention to treat analysis including all eligible participants who took at least one dose of study drug and had a least one follow-up AUA Symptom Score measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Saw Palmetto: One, two, and then three 320 mg gelcaps with dose escalations at 24 and 48 weeks.
- Placebo: One, two, and then three 320 mg placebo gelcaps with dose escalations at 24 and 48 weeks.
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -2.20 (5.83) [-3.04 to -0.36] | -2.99 (5.65) [-3.81 to -2.17]

2. Secondary Outcome: Participants Global Assessments of Improvement and Satisfaction at End of Study.
Description: Participants' global assessments of improvement and satisfaction at the end of the study. Likert scales were transformed to a 0 - 100 scale. The lowest possible score is 0 and the highest possible score is 100, which would reflect better outcomes.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale
  Global Assessment: Change from Baseline | 49.9 (26.9) [46.0 to 54.0] | 50.58 (28.7) [46.0 to 55.0]
  Global Assessment: Satisfaction with Symptoms | 48.9 (26.9) [44.9 to 52.9] | 50.6 (28.8) [46.4 to 54.8]

3. Secondary Outcome: Benign Prostate Hyperplasia (BPH) Impact Index Score
Description: The mean difference in the BPH Impact Index score from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The BPH Index Score is a self administered 4 item index. Three questions are scored on a scale from 0 to 3, with zero being none, one being only a little, two being some, and three being a lot. One question is scored on a scale from 0 to 4, with zero being none of the time, one being a little of the time, two being some of the time, three being most of the time, and four being all of the time. The lowest possible score is 0 and the highest possible score is 13, which would represent the greatest dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.81 (2.38) [-1.16 to -0.46] | -1.23 (2.57) [-1.60 to -0.87]

4. Secondary Outcome: International Prostate Symptom Score Quality of Life (IPSS QOL) Score
Description: The mean difference in the IPSS Quality-of-Life Question from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The IPSS Quality-of-Life Question is an additional question to the AUA Symptom Score. The self administered question is scored on a scale from 0 to 6, with zero being delighted, one being pleased, two being mostly satisfied, three being mixed-about equally satisfied and dissatisfied, four being mostly dissatisfied, five being unhappy, and six being terrible. The lowest possible score is 0 and the highest possible score is 6, which would represent the greatest dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.34 (1.26) [-0.52 to -0.16] | -0.49 (1.27) [-0.67 to -0.31]

5. Secondary Outcome: American Urological Association(AUA) Nocturia Item
Description: The mean difference in the nocturia item of the AUA Symptom Score from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The nocturia item is a self administered question from the AUA Symptom Score Index that assesses the number of times a participant typically gets up to urinate from the time he goes to bed at night until the time he gets up in the morning. The question is scored on a scale of zero to five, with zero being none, one being one time, two being two times, three being three times, four being four times, and five being five or more times. The lowest possible score is 0 and the highest possible score is 5, which would represent the highest level dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.36 (1.22) [-0.72 to 0] | -0.15 (1.22) [-0.44 to 0.13]

6. Secondary Outcome: Peak Uroflow
Description: The mean difference in the participants' peak uroflow from baseline to 72 weeks in the modified intention to treat analysis. The peak uroflow was measured in milliliters/seconds. The higher units indicated greater dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/sec
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
mL/sec | -0.18 (6.03) [-1.07 to .70] | -0.79 (5.55) [-1.58 to 0]

7. Secondary Outcome: Post-void Residual
Description: The mean difference in the participants' post-void residual from baseline to 72 weeks in the modified intention to treat analysis. The post-void residual was measured in milliliters. The higher units indicated greater dysfunction.
Time Frame: Baseline to 72 weeks
Population: The analysis population was determined by the number of participants that were randomized and included in the modified intention to treat analyses.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
mL | 4.78 (83.70) [-30.00 to 52] | 1.17 (76.12) [-33.00 to 34]

8. Secondary Outcome: Prostate Specific Antigen (PSA) Level
Description: The mean difference in the PSA level from baseline to 72 weeks in the modified intention to treat analysis. The PSA level was measured in nanograms/milliliters. The higher units indicated greater dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
ng/mL | 0.32 (0.82) [-0.08 to 0.73] | -0.19 (1.16) [-0.53 to 0.14]

9. Secondary Outcome: International Index of Erectile Function (IIEF)Scale Score.
Description: The mean difference in the IIEF score from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The IIEF is a multidimensional scale for assessment of erectile dysfunction. The six item self administered questionnaire is scored on a scale from 0 to 5, with zero being no sexual activity, one being never or almost never, two being a few times (much less than half the time), three being sometimes (much less than half the time), four being most times (much more than half the time), and five being always or almost always. The lowest possible score is 0 and the highest possible score is 30, which represents less dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.52 (7.59) [-1.63 to 0.59] | -1.06 (7.39) [-2.11 to -0.02]

10. Secondary Outcome: Male Sexual Health Questionnaire - Ejaculatory Domain (MSHQ-EjD) Scale Score.
Description: The mean difference in the MSHQ-EjD from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The MSHQ-EjD scale is used for the assessment ejaculatory dysfunction (EjD). The MSHQ-EjD consists of four self administered questions. Three of the items are scored on a scale from 0 to 5, with zero being all the time, one being most of the time, two being some of the time, three being a little of the time, four being none of the time, and five being no sexual activity. The fourth item is scored on a scale of 1 - 5, with one being not at all bothered, two being a little bit bothered, three being moderately bothered, four being very bothered, and five being extremely bothered. The lowest possible score is 0 and the highest possible score is 20, which represents the highest level of dysfunction.
Time Frame: Baseline to 72 weeks.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.38 (4.51) [-1.04 to 0.28] | -0.09 (3.75) [-0.63 to 0.45]

11. Secondary Outcome: International Continence Society Male Incontinence Symptom (ICSmale IS) Score
Description: The mean difference in the ICSmaleIS score from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The six item self administered questionnaire is scored on a scale from 0 to 4, with zero being never, one being occasionally, two being sometimes, three being most of the time, and four being all of the time. The lowest possible is 0 and the highest possible score is 24, which represents the the highest level of dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.48 (2.22) [-0.80 to -0.16] | -0.84 (2.46) [-1.17 to -0.51]

12. Secondary Outcome: Jenkins Sleep Scale Score
Description: The mean difference in the Jenkins Sleep Dysfunction score from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. Jenkins Sleep Dysfunction score is used to assess sleep dysfunction. The four item self administered questionnaire is scored on a scale from 0 to 5, with zero being not at all, one being 1 -3 days, two being 4 - 7 days, three being 8 - 14 days, four being 15 - 21 days, and five being 22 - 31 days. The lowest possible score is 0 and the highest possible score is 20, which represents the highest level of dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.80 (3.59) [-1.34 to -0.27] | -1.63 (4.38) [-2.25 to -1.01]

13. Secondary Outcome: NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Pain Scale
Description: The mean difference in the NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Pain Scale score from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Pain Scale is a four item self administered questionnaire. Three of the four items are scored on a scale from 0 - 1, with zero being no and one being yes. The fourth item is scored on a scale from 0 - 10, with zero being no pain and ten being pain as bad as you can imagine. The lowest possible score is 0 and the highest possible score is 21, which represents the highest level of pain.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | 0 (2.85) [-0.08 to 0] | 0 (2.82) [-1.00 to 0]

14. Secondary Outcome: NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Urinary Symptom Scale
Description: The mean difference in the NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) urinary symptom scale from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) urinary symptom scale consists of two self administered questions. The questions are scored on a scale from 0 - 5, with zero being not at all, one being less than 1 time in 5, two being less than half the time, three being about half the time, four being more than half the time, and five being almost always. The lowest possible score is 0 and the highest possible score is 10, which represents the highest level of dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.35 (2.19) [-0.67 to -0.03] | -0.86 (2.53) [-1.22 to -0.49]

15. Secondary Outcome: NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Quality of Life (QOL)Scale
Description: The mean difference in the NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Quality of Life (QOL) scale from baseline to 72 weeks in participants that were included in the modified intention to treat analysis. The NIH-Chronic Prostatitis Symptom Index (NIH-CPSI) Quality of Life (QOL) scale consists of three self administered questions. Two of the questions are scored on a scale of 0 - 3, with zero being none, one being only a little, two being some, and three being a lot. The third question is scored on a scale of 0 -6, with zero being delighted, one being pleased, two being mostly satisfied, three being mixed (equally satisfied and dissatisfied), four being mostly dissatisfied, five being unhappy, and six being terrible. The lowest possible score is 0 and the highest possible score is 12, which represents the highest level of dysfunction.
Time Frame: Baseline to 72 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Saw Palmetto | Placebo
Number analyzed (Participants) | 176 | 181
units on a scale | -0.85 (2.14) [-1.16 to -0.53] | -1.08 (2.16) [-1.39 to -0.77]

ADVERSE EVENTS:
Time Frame: Collected over 72 weeks
Description: The number of participants at risk was determined by the number of participants that were randomized and included in the modified intention to treat analyses.
Arm/Group | Saw Palmetto | Placebo
Serious Adverse Events (participants affected / at risk) | 18/176 | 17/181
Other Adverse Events (participants affected / at risk) | 138/176 | 139/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saw Palmetto (N=176) | Placebo (N=181)
Appendectomy for appendicitis (Surgical and medical procedures) | 0 (0) | 1 (1)
Appendectomy for ruptured appendix (Surgical and medical procedures) | 0 (0) | 1 (1)
Automobile accident with multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back surgery for a lumbar spinal connective tissue cyst (Surgical and medical procedures) | 0 (0) | 1 (1)
Bacterial epididymitis requiring intravenous antibiotics (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Colon resection for a polyp (Surgical and medical procedures) | 0 (0) | 1 (1)
Elective knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Elective plastic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective repair of abdominal aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Elective tonsillectomy and deviated nasal septum repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Episode of atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Gross hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospitalized after pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalized for abdominal pain, underwent laparascopic cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalized for cellulitis of the elbow, required intravenous antibiotics (Infections and infestations) | 0 (0) | 1 (1)
Hospitalized for chest pain (General disorders) | 0 (0) | 1 (1)
Hospitalized for chest pain due to coronary artery disease, underwent revascularization (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalized for chest pain that proved noncardiac after the study (General disorders) | 0 (0) | 1 (1)
Hospitalized for diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Hospitalized for hypotension due to pneumonia and chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospitalized for knee pain secondary to torn vastus lateralis muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hospitalized for pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hospitalized for radioactive iodine treatment for thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Inferior wall myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Lower gastointestinal diverticular bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mestatic recurrent follicular thyroid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sepsis secondary to a pelvic fracture (Infections and infestations) | 1 (1) | 0 (0)
Severe Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Small bowel obstruction requiring laparoscopy lysis of adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope with transient high grade atrioventricular block (Nervous system disorders) | 1 (1) | 0 (0)
Upper gastrointestinal bleeding requiring transfusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saw Palmetto (N=176) | Placebo (N=181)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Cold (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 19 (19)
Frost bite to bronchial tubes (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increase mucus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Strep Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (12)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (10)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Post Nasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pre-Existing Lower Back Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsilectomy and Deviated Septum Repair (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 13 (13)
Knee Pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (8)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10)
Elbow Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Broken Tooth (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest Discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hernia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Facial Edema (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
C-Spine Degenerative Disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruised Ribs/Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fore Arm Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Lump in Right Calf (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hand Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Toe Surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee Replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sciatic Nerve Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Sore Coccyx (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wrist Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 10 (10) | 7 (7)
Decreased Libido (Renal and urinary disorders) | 3 (3) | 3 (3)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 4 (4)
Elevated PSA (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular Pain (Renal and urinary disorders) | 2 (2) | 2 (2)
Tip of Penis Swollen (Renal and urinary disorders) | 2 (2) | 0 (0)
BPH Symptoms (Renal and urinary disorders) | 27 (27) | 33 (33)
Pain in Groin (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 3 (3) | 2 (2)
Prostatitis (Renal and urinary disorders) | 2 (2) | 2 (2)
Small Spermatocele found in physical exam (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostate nodule left lobe (Renal and urinary disorders) | 1 (1) | 0 (0)
Peyronies Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Increase Firmness Erection (Renal and urinary disorders) | 1 (1) | 0 (0)
Anal Itching (Renal and urinary disorders) | 0 (0) | 1 (1)
Epididymitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Increased PVR (Renal and urinary disorders) | 0 (0) | 1 (1)
Trace WBC in Urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Urological Disorder - Bloating (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (7)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Reflux (Gastrointestinal disorders) | 4 (4) | 5 (5)
Abdominal Pains (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal Bleed (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Barrett's Esophagus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Fatty Liver (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
White Stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upset Stomach/Flu (Gastrointestinal disorders) | 1 (1) | 9 (9)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Black Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon Polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Itching (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes